CLINICAL TRIAL: NCT00848341
Title: Canadian Registry of ICD Implant Testing Procedures
Status: Completed | Type: Observational
Sponsor: Guidant Corporation (Industry)
Responsible Party: Dr Jeff Healey, hamilton health sciences center
Other Study IDs: CREDIT
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Ventricular Fibrillation
MeSH Terms: conditions — Ventricular Fibrillation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Control
  Interventions: Device: GUIDANT ICD SYSTEM

INTERVENTIONS:
Device: GUIDANT ICD SYSTEM

SUMMARY:
To document practices in Canadian ICD implant centres around defibrillation therapy efficacy testing.

DETAILED DESCRIPTION:
To document types of defibrillation testing (DFT) procedures are in current use in Canada, rates of use an dno use of DFT testing, medical indications for non use of DFT testing, rate of successful testing of first lead configuration, rates and types of complications from DFT testing, costs of implant procedures and the costs associated with DFT testing, short term outcomes of patients with different types of implant procedures.

ELIGIBILITY:
Inclusion Criteria:

* Receiving a Guidant ICD system, including replacements

Exclusion Criteria:

* New epicardial lead(s) implanted, included in another cardiovascular trial (may be in the ELECTION Study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who are indicated for a market approved ICD
Sampling Method: Non-Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2006-01; Primary Completion 2008-04 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
to systematically collect and quanitfy characteristics of ICD implant procedures in Canadian Hospitals | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Connolly, MD, Principal Investigator — Hamilton Health Sciences Center